CLINICAL TRIAL: NCT07150884
Title: A Randomized, Double-blind, Patient-control Trial to Study Weight Gain in Premature Newborns Receiving Lactase-fortified Milk
Brief Title: Lactase-Assisted Control Trial On Weight GAin in INfants.
Acronym: LACTOGAIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Dimitrios Rallis, Assistant Professor in Pediatrics and Neonatology, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 701/22-01-2025
Record Dates: First submitted 2025-08-27; First posted 2025-09-02 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-08

CONDITIONS: Premature - Weight 1000g-2499g or Gestation of 28-37weeks; Healthy
Keywords: Lactase; Prematurity; Human milk; Weight gain; Feeding intolerance
MeSH Terms: conditions — Premature Birth; Weight Gain | interventions — Lactase

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lactase-Fortified Milk (Experimental): Newborns in the lactase group will receive milk fortified with 2 drops of lactase/kg of body weight per meal. The enrichment of the milk with lactase drops will be carried out by the nurse on duty without it being known by the principal investigator to which group (lactase group or control group) each newborn belongs. Only a secondary researcher and the shift nurse will have access to neonatal randomization information.
  The lactase drops that will be used in the study will be Delictase®, which is a dietary supplement that helps the proper digestion of lactose through its breakdown. Delictase® lactase drops offer an exogenous source of the lactase enzyme, which is essential for the proper absorption and digestion of lactose, can be administered from birth, mixed into the administered milk and contain high levels of lactase (>3,000 ALU*). The supply of Delictase® lactase preparations will be carried out by Galenic Pharmacy, every 2 months at the study site.
  Interventions: Dietary Supplement: Lactase
- Control (No Intervention): The feeding of the newborns of the study will be in accordance with the usual practices of the clinic, i.e. the first choice will be breast milk, the second the human milk of the donor from the milk bank and the third choice the formula of premature newborns. Breast milk boosters will be added to breast milk according to the usual clinic practices, i.e. when the volume of milk administered exceeds 25 ml per meal.
  Human milk is given an estimated caloric value of 68 kcal/100 mL, while premature formula is given 81 kcal/100 mL.

INTERVENTIONS:
Dietary Supplement: Lactase — The lactase drops that will be used in the study will be Delictase®, which is a dietary supplement that helps the proper digestion of lactose through its breakdown. Delictase® lactase drops offer an exogenous source of the lactase enzyme, which is essential for the proper absorption and digestion of lactose, can be administered from birth, mixed into the administered milk and contain high levels of lactase (>3,000 ALU*). The supply of Delictase® lactase preparations will be carried out by Galenic Pharmacy, every 2 months at the study site.
  Arms: Lactase-Fortified Milk

SUMMARY:
Lactose, a disaccharide that includes the monosaccharides glucose and galactose, is the main carbohydrate found exclusively in mammalian milk. Lactase is found in the intestinal mucosa and is located at the ends of the villi, while it is a factor of maximum clinical importance in milk tolerance and in the occurrence of diarrheal disease. Developmental lactase deficiency is defined as the relative lactase deficiency observed in premature newborns less than 34 weeks of gestation. In the immature gastrointestinal tract, lactase and other disaccharidas are deficient until at least 34 weeks of gestation. One study in premature babies reported a benefit from the use of lactase-supplemented or lactose-reduced formulas, while the use of lactose-containing formulas and human milk did not appear to have short- or long-term harmful effects on infants and infants. Up to 20% of dietary lactose can reach the colon in newborns and young infants.

Due to the inadequate functional development of lactase, premature infants may not digest and absorb the main source of carbohydrate energy, lactose. The high osmotic load associated with indigestible lactose is one of the many possible causes of diarrhea and food intolerance in premature babies. As a result of diarrhea stools and small bowel damage, the already low functional activity of lactase will be further reduced affecting weight gain, while it takes up to 2 weeks for lactase activity to be restored.

Carlson et al showed that the addition of lactase to premature formula reduces the amount of lactose by 70%, with a negligible effect on osmolarity. Previous studies have found that premature infants fed a reduced lactose formula had a better weight gain rate than those who took 100% lactose formula. In two of these studies, weight gain improved despite eating fewer calories.

In the present study we intend to test whether the use of lactase to hydrolysis lactose in premature milk would result in better weight gain and improved dietary tolerance by taking the same calorie intake. This is a prospective, double-blind, randomized study to evaluate tolerance and weight gain in premature infants who received either (1) human milk or premature formula enriched with Delictase ® drops (lactase group) or (2) unfortified human milk or premature formula (control group).

The study will be carried out at the Second Neonatal Clinic and Neonatal Intensive Care Unit of the Aristotle University of Thessaloniki, in premature newborns (gestational age [GA] 28-34 weeks) who will be hospitalized in the Neonatal Intensive Care Unit.

The study will enroll newborns (1) with a gestational duration of 28 to 34 weeks, (2) who receive ≥75% of their energy needs intestinally, (3) with the absence of severe congenital malformations or gastrointestinal diseases, including necrotizing enterocolitis (NEC) (4) without taking postnatal steroids or diuretics. Small, suitable and large for newborns of gestational age will be eligible for the study.

Exclusion criteria will be neonates whose guardians refuse to participate in the study, neonates with congenital malformations or gastrointestinal diseases, and neonates receiving postnatal steroids or diuretics.

The participation of newborns in the study will take place after written consent of the parents after information.

DETAILED DESCRIPTION:
Lactose, a disaccharide that includes the monosaccharides glucose and galactose, is the main carbohydrate found exclusively in mammalian milk. The absorption of lactose requires lactase activity to break the bond that binds the 2 monosaccharides. Lactase is found in the intestinal mucosa and is located at the ends of the villi, while it is a factor of maximum clinical importance in milk tolerance and in the occurrence of diarrheal disease.

Milk intolerance can be attributed to either lactose or protein content. Lactose intolerance may occur in infants and young children with acute diarrhoea, although its clinical significance is limited. Lactose intolerance symptoms are relatively common among older children and adolescents. However, associated intestinal damage is rarely observed. Lactose tolerance is a separate entity from cow's milk protein allergy, which is of immune etiology and can cause varying degrees of intestinal mucosal injury. Cow's milk protein intolerance is reported in 2% to 5% of infants within the first 1 to 3 months of life, usually subsides by the age of 1 year and is not the subject of this statement.

In more specific cases, the hydrogen breath test is the least invasive and most helpful test for diagnosing lactose malabsorption. The test is performed by administering a standardized amount of lactose (2 g/kg, up to a maximum of 25 g, equivalent to the amount of lactose in 2 glasses of milk) after fasting overnight and then measuring the amount of hydrogen in the exhaled air for a period of 2 to 3 hours. An increase (20 ppm) in hydrogen after about 60 minutes is indicative of lactose malabsorption. Factors that may produce false negative or false positive results include conditions affecting the intestinal flora (e.g., recent use of antimicrobial agents), lack of hydrogen-producing bacteria (10%-15% of the population), ingestion of a high-fiber diet before testing, bacterial overgrowth of the small intestine, or intestinal motility disorders.

In newborns and infants with diarrhea in whom lactose (or other carbohydrate) intolerance is suspected, the stool can be checked for carbohydrate malabsorption by testing the pH of the stool, which is reduced by carbohydrate malabsorption as a result of the formation of volatile fatty acids. It is noted that the pH of the stool is lower in infants compared to older children and adolescents due to the normal overload of lactose in their diet; which in turn helps to promote the growth of Lactobacillus species in the large intestine. Reducing substances can also be detected in the stool, such as reducing sugars that include lactose, glucose, fructose and galactose, but not sucrose. Because some patients may only absorb enough carbohydrates, such as lactose, to lower the pH of the stool but not increase the excretion of carbohydrates in the stool, the pH test is a more sensitive test for carbohydrate malabsorption.

Developmental lactase deficiency is defined as the relative lactase deficiency observed in premature newborns less than 34 weeks of gestation. In the immature gastrointestinal tract, lactase and other disaccharidesas are deficient until at least 34 weeks of gestation. One study in premature babies reported a benefit from the use of lactase-supplemented foods or lactose-reduced preparations. While the use of lactose-containing preparations and human milk does not appear to have short- or long-term harmful effects on newborns and infants. Up to 20% of dietary lactose can reach the colon in newborns and young infants. The metabolism of lactose by colon microbes lowers the pH of the stool, which has a beneficial effect, favoring certain organisms (e.g. Bifidobacterium and Lactobacillus species) instead of potential pathogens (Proteus, Escherichia coli and Klebsiella species) in young infants.

Lactase is detected for the first time in the fetus from the 10th week of gestation. At 28 to 34 weeks, lactase activity is only ~30% of that found at the end of pregnancy. At 35 to 38 weeks, it reaches 70% of the activity of the end months. Due to the inadequate functional development of lactase, premature infants may not digest and absorb the main source of carbohydrate energy, lactose. The high osmotic load associated with indigestible lactose is one of the many possible causes of diarrhea and food intolerance in premature babies. As a result of diarrhea stools and small bowel damage, the already low functional activity of lactase will be further reduced affecting weight gain, while it takes up to 2 weeks for lactase activity to be restored.

Lactose intolerance is often treated with soy proteins, protein hydrolysis products, low-lactose, or lactose-free formulas. However, these types do not meet the nutritional requirements for the development and development of premature newborns, which need human milk with a human milk booster or premature milk. Ideally, premature babies with lactose intolerance should take these hydrolyzed lactose foods. Carlson et al showed that the addition of lactase to premature formula reduces the amount of lactose by 70% after a 2-hour incubation period at room temperature, with negligible effect on osmolarity. Previous studies have found that premature infants fed a reduced lactose formula had a better weight gain rate than those who took 100% lactose formula. In two of these studies, weight gain improved despite eating fewer calories.

In the present study we intend to test whether the use of lactase to hydrolysis lactose in premature milk would result in better weight gain and improved dietary tolerance by taking the same calorie intake.

METHOD Study Population A prospective, double-blind, randomized study will be conducted to evaluate tolerance and weight gain in premature infants who received either (1) human milk or premature formula fortified with Delictase ® drops (lactase group) or (2) unfortified human milk or premature formula (control group).

Study Day 1 will be the day on which intestinal feeding will provide ≥75% of the daily intake of caloric needs. The study will be terminated when the newborn reaches 36 weeks or is discharged from the unit, whichever comes first.

Inclusion criteria The study will enrol newborns (1) with a gestational duration of 28 to 34 weeks, (2) who receive ≥75% of their energy needs intestinally, (3) with the absence of severe congenital malformations or gastrointestinal diseases, including necrotizing enterocolitis (NEC) (4) without taking postnatal steroids or diuretics. Small, suitable and large for newborns of gestational age will be eligible for the study.

Exclusion criteria Exclusion criteria will be neonates whose guardians refuse to participate in the study, neonates with congenital malformations or gastrointestinal diseases, and neonates receiving postnatal steroids or diuretics.

Feeding newborns The feeding of the newborns of the study will be in accordance with the usual practices of the clinic, i.e. the first choice will be breast milk, the second the human milk of the donor from the milk bank and the third choice the formula of premature newborns. Breast milk boosters will be added to breast milk according to the usual clinic practices, i.e. when the volume of milk administered exceeds 25 ml per meal.

Human milk is given an estimated caloric value of 68 kcal/100 mL, while premature formula is given 81 kcal/100 mL.

Randomization Guardians of newborns who meet the criteria for inclusion in the study will be approached to be informed about participation in the study. Newborns whose guardians consent to participate will be included in the study.

Newborns, after enrolment in the study, will be randomized to either the lactase group or the control group. The results of randomization will not be known to the principal investigator until after the study is completed.

Intervention Newborns in the lactase group will receive milk fortified with 2 drops of lactase/kg of body weight per meal. The enrichment of the milk with lactase drops will be carried out by the nurse on duty without it being known by the principal investigator to which group (lactase group or control group) each newborn belongs. Only a secondary researcher and the shift nurse will have access to neonatal randomization information.

The lactase drops that will be used in the study will be Delictase®, which is a dietary supplement that helps the proper digestion of lactose through its breakdown. Delictase® lactase drops offer an exogenous source of the lactase enzyme, which is essential for the proper absorption and digestion of lactose, can be administered from birth, mixed into the administered milk and contain high levels of lactase (>3,000 ALU*). The supply of Delictase® lactase preparations will be carried out by Galenic Pharmacy, every 2 months at the study site.

Recording of results For all newborns in the study, perinatal and neonatal data will be recorded on computers anonymously by the researchers. Somatometric data (body weight, head circumference, body length) will be recorded at birth and per week until the completion of the study. Biochemical markers of homeostasis (Your, Cr, Proteins, Albumin, Na, K, Ca, P, Mg, AST, ALT, ALP, TG, Cholesterol, HDL, LDL) will also be recorded according to the usual practices of neonatal hospitalization in the NICU. Caloric intake and type of food will be recorded daily The main outcome variable will be weight gain (g/day). Additional outcome variables included benefits in body length and head circumference (cm/week). Also the concentrations of protein, albumin, sodium and potassium in the serum. and measurements of feeding tolerance (vomiting, gastric residual tumors, stool count, and stool reductives) will be recorded. Finally, any withdrawal from the study due to food intolerance or NEC will be recorded.

Statistical analysis According to previous studies, the main outcome of the study (weight gain, g/day) was used as the basis for calculating the sample size. A total of 100 newborns (50 newborns per group) allows the detection of a 33% increase in mean weight gain per day in the treatment group, with a strength of 0.80. The differences between the groups are considered statistically significant at the level of P <.05.

Neonatal characteristics of the lactase and control group will be compared with the t-test in terms of continuous variables (caloric intake, weight gain, length, head circumference, gastric residual volume, daily number of vomiting episodes, daily stool count, and serum albumin, total protein, sodium, and potassium concentrations) or the Mann-Whitney test for variables with abnormal dispersion. The Pearson X2 or Fisher exact test will be used to compare the categorical variables (proportion of neonates in each group who developed food intolerance, had at least one episode of vomiting during the study, withdrew from the study due to medical condition or parental request, or experienced NEC) between the two groups.

Retrograde analysis will be used to check the correlation of weight gain with lactase administration or not, stratified for perinatal and neonatal factors with statistical significance.

Duration of the study Recruitment is expected to begin in August 2025 and be completed within 24 months.

ELIGIBILITY:
Inclusion Criteria:

The study will enrol newborns (1) with a gestational duration of 28 to 34 weeks, (2) who receive ≥75% of their energy needs intestinally, (3) with the absence of severe congenital malformations or gastrointestinal diseases, including necrotizing enterocolitis (NEC) (4) without taking postnatal steroids or diuretics. Small, suitable and large for newborns of gestational age will be eligible for the study.

Exclusion Criteria:

Exclusion criteria will be neonates whose guardians refuse to participate in the study, neonates with congenital malformations or gastrointestinal diseases, and neonates receiving postnatal steroids or diuretics.

Ages: 1 Day to 4 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2025-08-27 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Weigh Gain | 2-4 weeks
  The main outcome variable will be weight gain (g/day).

SECONDARY OUTCOMES:
Body length | 2-4 weeks
  Benefits in body length (cm/week).
Head circumference | 2-4 weeks
  Benefits in head circumference (cm/week).

OTHER OUTCOMES:
Biochemistry | 2-4 weeks
  The concentrations of protein, albumin, sodium and potassium in the serum will be recorded
Feeding intolerance | 2-4 weeks
  Measurements of feeding tolerance (vomiting, gastric residual tumors, stool count, and stool reductives) will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Christos Tsakalidis, Study Director — Aristotle University Of Thessaloniki
Locations (1):
- Papageorgiou General Hospital, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shulman RJ, Feste A, Ou C. Absorption of lactose, glucose polymers, or combination in premature infants. J Pediatr. 1995 Oct;127(4):626-31. doi: 10.1016/s0022-3476(95)70128-1. PMID 7562290
- [Background] Kien CL, McClead RE, Cordero L Jr. Effects of lactose intake on lactose digestion and colonic fermentation in preterm infants. J Pediatr. 1998 Sep;133(3):401-5. doi: 10.1016/s0022-3476(98)70278-1. PMID 9738725
- [Background] Kien CL, Liechty EA, Mullett MD. Effects of lactose intake on nutritional status in premature infants. J Pediatr. 1990 Mar;116(3):446-9. doi: 10.1016/s0022-3476(05)82842-2. No abstract available. PMID 2308040
- [Background] Griffin MP, Hansen JW. Can the elimination of lactose from formula improve feeding tolerance in premature infants? J Pediatr. 1999 Nov;135(5):587-92. doi: 10.1016/s0022-3476(99)70057-0. PMID 10547247
- [Background] Meetze WH, Valentine C, McGuigan JE, Conlon M, Sacks N, Neu J. Gastrointestinal priming prior to full enteral nutrition in very low birth weight infants. J Pediatr Gastroenterol Nutr. 1992 Aug;15(2):163-70. doi: 10.1097/00005176-199208000-00011. PMID 1403464
- [Background] Reis BB, Hall RT, Schanler RJ, Berseth CL, Chan G, Ernst JA, Lemons J, Adamkin D, Baggs G, O'Connor D. Enhanced growth of preterm infants fed a new powdered human milk fortifier: A randomized, controlled trial. Pediatrics. 2000 Sep;106(3):581-8. doi: 10.1542/peds.106.3.581. PMID 10969106
- [Background] Schanler RJ. The low-birth weight infant. In: Walker WA, Watkins JB, eds. Nutrition in pediatrics: basic science and clinical application. 2nd ed. Hamilton, Ontario, Canada: BC Decker Inc; 1996. p. 392-412.
- [Background] American Academy of Pediatrics Com- mittee on Nutrition. Pediatric Nutrition Handbook. 4th ed. Elk Grove (IL): American Academy of Pediatrics; 1998. p. 69
- [Background] Nutrition Committee of the Canadian Pediatric Society. Nutrient needs and feeding of preterm infants. Can Med Assoc J 1995;52:1756-85.
- [Background] Sinden AA, Sutphen JL. Dietary treatment of lactose intolerance in infants and children. J Am Diet Assoc. 1991 Dec;91(12):1567-71. PMID 1960350
- [Background] Carlson SJ, Rogers RR, Lombard KA. Effect of a lactase preparation on lactose content and osmolality of preterm and term infant formulas. JPEN J Parenter Enteral Nutr. 1991 Sep-Oct;15(5):564-6. doi: 10.1177/0148607191015005564. PMID 1942472
- [Background] Lebenthal E, Lee PC, Heitlinger LA. Impact of development of the gastrointestinal tract on infant feeding. J Pediatr. 1983 Jan;102(1):1-9. doi: 10.1016/s0022-3476(83)80276-5. PMID 6401326
- [Background] Brady MS, Rickard KA, Fitzgerald JF, Lemons JA. Specialized formulas and feedings for infants with malabsorption or formula intolerance. J Am Diet Assoc. 1986 Feb;86(2):191-200. PMID 3511129
- [Background] Saavedra JM, Perman JA. Current concepts in lactose malabsorption and intolerance. Annu Rev Nutr. 1989;9:475-502. doi: 10.1146/annurev.nu.09.070189.002355. No abstract available. PMID 2669882
- [Background] Kien CL. Carbohydrates. In: Tsang RC, Lucas A, Uauy R, et al, eds. Nu- tritional needs of the preterm infant: scientific basis and practical guide- lines. Baltimore (MD): Williams and Wilkins; 1993. p. 47-63.
- [Background] Groh-Wargo S. Gastrointestinal development. In: Groh-Wargo S, Thompson M, Hovasi Cox J, Hartline JV, editors. Nutritional care for high risk newborns. Chicago: Precept Press; 2000. p. 209-30.